CLINICAL TRIAL: NCT05842434
Title: Pilot Study of the Felix System in Patients With Essential Tremor and Parkinson's Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fasikl Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-1
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Essential Tremor; Parkinson Disease
MeSH Terms: conditions — Essential Tremor; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Felix (Experimental)
  Interventions: Device: Felix

INTERVENTIONS:
Device: Felix — Felix is a wrist-worn, noninvasive, transcutaneous neurostimulation system intended for daily use to suppress hand tremors. An artificial intelligence (AI) algorithm will automatically adjust the stimulation based on each patient's tremor throughout the day.

SUMMARY:
A prospective, open-label, multi-center pilot study designed to evaluate the safety and effectiveness of the Felix system in the relief of upper limb tremors in adults with essential tremor and Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Willing to provide written, informed consent to participate in the study.
3. For subjects with essential tremor (ET):

   1. A clinical diagnosis of ET.
   2. For either upper limb, a tremor severity score of 2 or higher as measured by one of the TETRAS items and a total score of 6 or higher across all TETRAS tasks.
4. For subjects with Parkinson's disease (PD):

   1. A clinical diagnosis of PD (MDS-PD criteria).
   2. A tremor score of 2 or higher on MDS-UPDRS question 3.15 (postural tremor) or 3.16 (kinetic tremor), OR
   3. A rest tremor score of 2 or higher on MDS-UPDRS question 3.17 (rest tremor amplitude) in one upper extremity and a score of 2 or higher on MDS-UPDRS question 3.18 (constancy of tremor).
5. Stable dosage of any medication, if applicable, for 30 days prior to study entry.
6. Familiar with operating a touch-screen smartphone and connecting to Wi-Fi internet at home.
7. If necessary, have a dedicated caregiver to help with study required activities, such as putting on the study device, etc.
8. Willing to comply with study protocol requirements including:

   1. Remaining on a stable dosage of current medications, if applicable, during the course of the study.
   2. Remaining on stable caffeine consumption, if applicable, during the course of t the study.
   3. No alcohol consumption on the day before a study visit.

Exclusion Criteria:

1. Prior limb amputation or any known symptomatic peripheral neuropathy condition of the involved upper extremity.
2. Any current drug or alcohol abuse.
3. Current unstable epileptic conditions with a seizure within 6 months of study entry.
4. Pregnant or nursing subjects and those who plan pregnancy during the course of the study.
5. Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin at the stimulation site.
6. Known allergy to adhesives.
7. History of Alzheimer's disease or dementia (Montreal Cognitive Assessment (MoCA)≤19).
8. Botulinum Toxin injection for hand tremor within 4 months prior to study enrollment.
9. Subject is currently participating or has participated in another interventional clinical trial in the last 30 days which may confound the results of this study, unless approved by the Sponsor.
10. Subject is unable to communicate with the investigator and staff.
11. Any health condition that in the investigator's opinion should preclude participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Tremor Research Group Essential Tremor Rating Assessment (TETRAS) Performance Subscale | Baseline to 7 days
  A subset of 6 performance tasks will be rated by a physician for each upper limb separately. Each task will be rated from 0 to 4, indicating the increasing severity of tremor.
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Baseline to 7 days
  Physician rated MDS-UPDRS Part III on a 5-point scale, from 0 (normal) to 4 (severe)
Clinical Global Impression of Severity (CGI-S) | Baseline to 7 days
  Physician rating on a 7-point scale, from 1 (normal) to 7 (amongst the most extreme tremor)
Clinical Global Impression of Improvement (CGI-I) | Baseline to 7 days
  Physician rating of tremor improvement on a 7-point scale, from 1 (very much improved) to 7 (very much worse)
Tremor Research Group Essential Tremor Rating Assessment (TETRAS) Activities of Daily Living (ADL) Subscale | Baseline to 7 days
  Patient rating on a 5-point scale, from 0 (normal) to 4 (severely abnormal)
Patient Global Impression of Severity (PGI-S) | Baseline to 7 days
  Patient rating on a 7-point scale, from 1 (normal) to 7 (amongst the most extreme tremor)
Patient Global Impression of Improvement (PGI-I) | Baseline to 7 days
  Patient rating of tremor improvement on a 7-point scale, from 1 (very much improved) to 7 (very much worse)
Tremor Power | Baseline to 7 days
  Assessed by device sensor.
Tremor Research Group Essential Tremor Rating Assessment (TETRAS) Modified Activities of Daily Living (mADL) Subscale | Baselinen to 7 days
  TETRAS mADL score is a composite sum of items 2 to 11 of the TETRAS ADL subscale and items 6 (bilateral) and 7 (dominant hand) of the TETRAS performance subscale (PS). TETRAS mADL score is calculated as the sum of all 12 items and ranges from 0 to 52.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Dewey III, MD, Principal Investigator — Parkinson's Disease and Movement Disorders Center of Boca Raton; Rajesh Pahwa, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Kansas Medical Center, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: No